CLINICAL TRIAL: NCT04503343
Title: Effects of Non-drug Therapy on Cognitive Function in Healthy Individuals and Patients With First Episode Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Jian-Jun Ou, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD201908
Record Dates: First submitted 2020-07-24; First posted 2020-08-07 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): subjects are randomly divided into the intervention group. and they will be given a one-time non-drug intervention(mindfulness training, relaxation training or electrical cerebellar stimulation).
  Interventions: Other: non-drug intervention
- control group (No Intervention): subjects are randomly divided into the control group and regularly followed up.

INTERVENTIONS:
Other: non-drug intervention — mindfulness training, relaxation training, or electrical cerebellar stimulation
  Arms: intervention group

SUMMARY:
Mindfulness training, relaxation training, and cerebellar electrical stimulation were used to intervene in the cognitive function of healthy individuals and individuals with first episode depression

DETAILED DESCRIPTION:
In this proposed study,the investigators will evaluate the effects of different non-pharmacological interventions (physical/psychological) on emotion-related cognitive function.This project will use a variety of intervention methods to conduct research in healthy individuals and patients with mood disorders. The main intervention methods include: (1) mindfulness training;(2) relaxation training;(3) cerebellar electrical stimulation.

The study will recruit 80 healthy subjects and 40 first-episode depression patients. The study consisted of three steps: First, subjects filled in personal data and completed the first screening, randomly assigned groups, and filled in the pre-intervention questionnaire;Second, give a one-time non-drug intervention (mindfulness training, relaxation training or cerebellar electrical stimulation);Step 3: After the intervention, the subjects filled in the post-intervention questionnaire and completed the cognitive task test.Clinical efficacy and safety assessment will be done at first time. The specific aims are to evaluate the effect of non-drug therapy on cognitive function in healthy individuals and patients with first episode depression. and the behavior was evaluated by cognitive function task.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy individuals group:

1. Aged between 16 and 34;
2. Does not meet the criteria of the DIAGNOSTIC and Statistical Manual of Mental Disorders, DSM-5,Does not meet the diagnosis of depression, bipolar disorder and other mental disorders.

First episode depression group:

1. Aged between 16 and 34;
2. Clinically diagnosed as having depression according to the DIAGNOSTIC and Statistical Manual of Mental Disorders (DSM-5);
3. First attack, not taking medicine, no risk of serious suicide NSSI.

Exclusion Criteria:

1. There are serious physical diseases, such as epilepsy, brain trauma, intracranial space-occupying lesions, severe audiovisual disorders, congenital heart disease, etc.;
2. Both Hamilton Depression Scale and Beck Depression Self-Rating Scale indicate severe depression or severe mental illness;
3. Affected by mental illness, it is difficult to conduct smooth and effective verbal communication and psychological measurement operation.

Ages: 16 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The change of mindfulness training on cognitive function in healthy individuals | baseline
  Cognitive function are measured by Faces Emotion Recognition Task
The change of mindfulness training on cognitive function in patients with first episode depression | baseline
  Cognitive function are measured by Emotional Categorisation Task
The change of cerebellar electrical stimulation on cognitive function in healthy individuals | baseline
  Cognitive function are measured by Emotional Recall Task

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Ou, doctor, Study Chair — Central South University; Runsen Chen, doctor, Study Director — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China